CLINICAL TRIAL: NCT04959734
Title: Impact of Covid-19 on Respiratory Syncytial Virus Seasonality and Disease Severity in UK Children (BronchStart)
Brief Title: COVID-19 Impact on RSV Emergency Presentations
Acronym: BronchSTART
Status: Recruiting | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Respiratory syncytial virus consortium in Europe (Unknown); Pediatric Emergency Research in the UK and Ireland (PERUKI) (Other)
Responsible Party: Sponsor
Other Study IDs: 140049
Record Dates: First submitted 2021-07-09; First posted 2021-07-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Bronchiolitis; Respiratory Syncytial Virus
Keywords: Bronchiolitis; RSV; Vaccine Effectiveness
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bronchiolitis: Infants less than 2 years who the clinician has diagnosed Bronchiolitis
- LRTI: Infants less than 2 years who the clinician has diagnosed a viral or bacterial lower respiratory tract infection
- Wheeze: Infants less than 2 years who the clinician has diagnosed the first presentation of a viral wheeze

SUMMARY:
Bronchiolitis is a very common winter disease that normally affects children less than one year of age. It is a common reason for parents and carers to bring their child to an Emergency Department (ED) and the frequent need for hospital admission means that paediatric units are at their capacity each winter.

During the COVID19 pandemic the virus that causes bronchiolitis (Respiratory Syncytial Virus; RSV) disappeared meaning this winter there have been virtually no cases of bronchiolitis in the United Kingdom. This phenomenon has been observed in many other countries around the world. Evidence from Australia suggests as restrictions such as social distancing for COVID19 are relaxed bronchiolitis returns, even in the summer. At the release of lockdown the return has been so dramatic in some areas of Australia the summer time numbers are above a typical winter. There is also evidence it may affect older children up to 2 years of age.

It is likely the Australian experience will be mirrored in the UK. The ability to track, anticipate and respond to a surge in bronchiolitis is important. There is a need to understand:

1. the onset of RSV spread at the earliest opportunity. This is important as some children are at higher risk of hospitalisation, intensive care admission or death if they contract RSV; knowing when to passively immunise these children is a public health priority.
2. whether the population at risk is a wider age range than normal and whether disease severity is greater as these will both effect service planning;

There are currently no existing studies or surveillance systems fully able to address these questions. This study will use staff in Emergency Department to report, in real time, case of bronchiolitis that they see and record essential, but non-identifying, information about them.

In 2022/23 the study evolved from a prospective surveillance study into a genomic analysis study with sites collecting positive respiratory samples for RSV genomic review.

In 2024/25 the study was amended in light of the introduction of the Bivalent Prefusion F Vaccine in Pregnancy in the United Kingdom to undertake a Vaccine Effectiveness study.

The main inclusion criteria remains the same but mothers who would have been eligible for the vaccine, and deliver an infant during the RSV season, were consented to obtain vaccination details so these could be linked to BronchSTART records.

ELIGIBILITY:
Inclusion Criteria:

i) Children under two years of age presenting to participating emergency departments with clinical features of:

* Bronchiolitis (cough, tachypnoea or chest recession, and wheeze or crackles on chest auscultation) or
* Lower Respiratory Tract infection or
* Afirst episode of acute viral wheeze.

Exclusion Criteria:

i) Children with previous episodes of wheeze responsive to bronchodilator (suggesting an underlying diagnosis of recurrent wheeze of early childhood)

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under two years of age attending emergency departments across the UK and Ireland
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Disposition | Confirmed at 7 Days following initial presentation
  Number of participants recorded via clinician or research nurse completed online case report form who are admitted or discharged from hospital following the initial presentation.
Intervention | Confirmed at 7 Days following initial presentation
  Rate of intervention in participants {Nasogastric Feed, Intravenous Fluids, Oxygen, High Flow Humidified Oxygen, CPAP or Mechanical Ventilation} determined by case note extraction and recorded by an online case report form up to 7 days following the initial presentation
Respiratory Syncytial Virus (RSV) Status | Confirmed at 7 Days following initial presentation
  Incidence of PCR confirmed RSV status (via PCR) if swabbed up to 7 days following the initial presentation

CONTACTS AND LOCATIONS:
Overall Officials: Damian Roland, BMBS PhD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Identifiable information is not collected as part of this study. The anonymised central database will be available on reasonable request.

REFERENCES:
- [Result] Williams TC, Marlow R, Hardelid P, Lyttle MD, Lewis KM, Mpamhanga CD, Cunningham S, Roland D; PERUKI. Clinical Impact of Serious Respiratory Disease in Children Under the Age of 2 Years During the 2021-2022 Bronchiolitis Season in England, Scotland, and Ireland. J Infect Dis. 2024 Jul 25;230(1):e111-e120. doi: 10.1093/infdis/jiad551. PMID 39052749
- [Result] Williams TC, Cunningham S, Drysdale SB, Groves H, Iskander D, Liu X, Lyttle MD, Marlow R, Maxwell-Hodkinson A, Mpamhanga CD, O'Hagan S, Sinha I, Swann OV, Waterfield T, Roland D; Paediatric Emergency Research in the UK and Ireland (PERUKI). Update to: Study Pre-protocol for "BronchStart - The Impact of the COVID-19 Pandemic on the Timing, Age and Severity of Respiratory Syncytial Virus (RSV) Emergency Presentations; a Multi-Centre Prospective Observational Cohort Study". Wellcome Open Res. 2024 Dec 18;6:120. doi: 10.12688/wellcomeopenres.16778.4. eCollection 2021. PMID 34458589
- [Result] Roland D, Williams T, Lyttle MD, Marlow R, Hardelid P, Sinha I, Swann O, Maxwell-Hodkinson A, Cunningham S. Features of the transposed seasonality of the 2021 RSV epidemic in the UK and Ireland: analysis of the first 10 000 patients. Arch Dis Child. 2022 Nov;107(11):1062-1063. doi: 10.1136/archdischild-2022-324241. Epub 2022 Sep 2. No abstract available. PMID 36261149